CLINICAL TRIAL: NCT05994833
Title: Virtual Physical Therapy Support for Runners Receiving Gait Analyses for Lower Body Running Related Musculoskeletal Issues
Brief Title: Virtual Physical Therapy Support for Runners
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB202301005
Record Dates: First submitted 2023-06-12; First posted 2023-08-16 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-02

CONDITIONS: Musculoskeletal Complication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- paper-based standard care exercise program (No Intervention)
- VPT (Experimental)
  Interventions: Behavioral: VPT

INTERVENTIONS:
Behavioral: VPT — The VPT will be comprised of weekly virtual visits with the participant for one month. During the visits, the physical therapist will review the exercises that were prescribed, adherence, provide feedback to the participant as they execute the exercises onscreen and make corrections, make any progression or adjustments to the exercises, review running cues they learned from the testing session and answer any questions. The therapist will also review any new activities that are initiated during the previous week (to control for confounders), changes in musculoskeletal pain and participation in running volume.
  Arms: VPT

SUMMARY:
This study will compare standard of care of home exercise for running rehabilitation to the combined treatment of home exercise with an individually provided four-session virtual physical therapy support program intervention on pain and physical function movements (controlled dual and single leg squat and lateral hopping in individuals post running injury. These collective findings will help provide new evidence of the responses to an individually provided virtual PT interventions among runners.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 to 65 years
* Regularly running at least 12 miles a week prior to development of musculoskeletal complaint.
* Free of surgical history of surgery to either lower limb
* No history of major bony injury to the lower limb such as traumatic fracture, within the past 12 months
* Presence of chronic lower body running related injuries (e.g., patellofemoral pain, IT band syndrome, Achilles tendinitis, chronic lower back pain after running)
* Body mass index (BMI) <=35 kg/m2

Exclusion Criteria:

* Pregnant women
* < 18 or 65 years
* BMI >35 kg/m2
* Mental disablement (down's syndrome or dementia)
* Any persons incarcerated, on parole, on probation, or awaiting trial.
* Individuals with neurologic or degenerative musculoskeletal disease, such as rheumatoid arthritis, muscular dystrophy, or Parkinson's disease.
* Current acute running related or sport related injury (e.g., ankle sprain, hip labral tear, ACL strain during an event or run)
* Individuals with a history of strong risk factors for poor fracture healing, such as uncontrolled diabetes, chemotherapy, end-stage organ disease, dialysis or smoking
* Unwilling to forgo your potential in-person therapy visits for a month after enrollment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2023-08-10 (Actual); Primary Completion 2029-08 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline numerical rating scale for pain (NRSpain) at 4 weeks | Visits 6; one month post enrollment
  A numerical rating scale for pain (NRSpain) will be used to assess changes in lower body related musculoskeletal pain at rest (now, average over the last week) and during weight bearing activity (like walking) on a range of lowest score of 0 (no pain) to 10 (worst pain)
Change from baseline numerical rating scale for pain (NRSpain) at 6 months | Visits 7; six months post enrollment
  A numerical rating scale for pain (NRSpain) will be used to assess changes in lower body related musculoskeletal pain at rest (now, average over the last week) and during weight bearing activity (like walking) on a range of lowest score of 0 (no pain) to 10 (worst pain)

SECONDARY OUTCOMES:
Change from baseline squat quality on single leg (using dominant leg) at 4 weeks | visit 6; one month post enrollment
  Squat performance on the single leg (using dominant leg) will be scored on a range of scale 1 (best performance) to 3 (worst performance)
Change from baseline squat quality on single leg (using dominant leg) at 6 months | visit 7; six months post enrollment
  Squat performance on the single leg (using dominant leg) will be scored on a range of scale 1 (best performance) to 3 (worst performance)
Change from baseline squat quality on the dual leg at 4 weeks | visit 6; one month post enrollment
  Squat performance on the dual leg will be scored on a range of scale 1 (best performance) to 3 (worst performance)
Change from baseline squat quality on the dual leg at 6 months | visit 7; six months post enrollment
  Squat performance on the dual leg will be scored on a range of scale 1 (best performance) to 3 (worst performance)
Change from baseline standing stork quality (using dominant leg) at 4 weeks | visit 6; one month post enrollment
  Balance performance on the standing stork will be scored on the ranges of excellent to poor scale compared to the normative data published for males/females (Schell & Leelarthaepin 1994)
Change from baseline standing stork quality (using dominant leg) at 6 months | visit 7; six months post enrollment
  Balance performance on the standing stork will be scored on the ranges of excellent to poor scale compared to the normative data published for males/females (Schell & Leelarthaepin 1994)
Change from baseline hopping quality (using dominant leg) at 4 weeks | visit 6; one month post enrollment
  Quality performance on the hopping three times (using dominant leg) and land on the same limb as far as possible will be scored based on the distance hopped, measured at the level of the great toe on a range of scale 1 (best performance) to 3 (worst performance)
Change from baseline hopping quality (using dominant leg) at 6 months | visit 7; six months post enrollment
  Quality performance on the hopping three times (using dominant leg) and land on the same limb as far as possible will be scored based on the distance hopped, measured at the level of the great toe on a range of scale 1 (best performance) to 3 (worst performance)
Change from baseline displacement in forward-backward direction during 20 sec of static standing position at 4 weeks | visit 6; one month post enrollment
  A markerless motion system will be used. Cameras will be used to collect the backward-forward displacement during 20 sec of static standing on both legs will be analyzed for ability to control static balance.
Change from baseline displacement in forward-backward direction during 20 sec of static standing position at 6 months | visit 7; six months post enrollment
  A markerless motion system will be used. Cameras will be used to collect the backward-forward displacement during 20 sec of static standing on both legs will be analyzed for ability to control static balance.
Change from baseline gait speed at 4 weeks | visit 6; one month post enrollment
  Spatiotemporal parameters are analyzed [i.e. gait speed (meters/sec), cadence (steps/minute)]
Change from baseline gait speed at 6 months | visit 7; six months post enrollment
  Spatiotemporal parameters are analyzed [i.e. gait speed (meters/sec), cadence (steps/minute)]
Change from baseline displacement of the center of gravity in vertical direction at 4 weeks | visit 6; one month post enrollment
  Spatiotemporal parameters are analyzed (i.e. center of gravity vertical displacement measured in centimeters)
Change from baseline displacement of the body in vertical direction at 6 months | visit 7; six months post enrollment
  Spatiotemporal parameters are analyzed (i.e. center of gravity vertical displacement measured in centimeters)
Change from baseline displacement between strides at 4 weeks | visit 6; one month post enrollment
  Spatiotemporal parameters are analyzed (i.e. stride width measured in centimeters)
Change from baseline displacement between strides at 6 months | visit 7; six months post enrollment
  Spatiotemporal parameters are analyzed (i.e. stride width measured in centimeters)

CONTACTS AND LOCATIONS:
Overall Officials: Sharareh Sharififar, PhD, PT, Principal Investigator — University of Florida
Locations (1):
- University of Florida College of medicine- Dept of PM&R, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No